CLINICAL TRIAL: NCT04540068
Title: Prediction of Transforaminal Epidural Injection Success in Sciatica
Brief Title: Prediction of TEI Success in Sciatica
Acronym: POTEISS
Status: Recruiting | Type: Observational
Sponsor: Eduard Verheijen (Other)
Collaborators: Spaarne Gasthuis (Other)
Responsible Party: Sponsor-Investigator, Eduard Verheijen, Bsc., Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Other Study IDs: POTEISS
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Radiculopathy; Lumbar Disc Herniation; Lumbar Spinal Stenosis
Keywords: Transforaminal Epidural Injection; Lumbar spine; Prospective cohort study; Prediction of success
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Lumbar Disc Herniation: Patients with a lumbar disc herniation on MRI and consistent with clinical findings are screened if they have an appointment at the pain clinic for treatment with a transforaminal epidural injection.
  Interventions: Drug: Transforaminal Epidural Injection
- Patients with Lumbar Spinal Stenosis: Patients with a lumbar spinal stenosis on MRI and consistent with clinical findings are screened if they have an appointment at the pain clinic for treatment with a transforaminal epidural injection.
  Interventions: Drug: Transforaminal Epidural Injection

INTERVENTIONS:
Drug: Transforaminal Epidural Injection — Injections above L3 will contain 1,5 ml lidocaine 1% and 10 mg dexamethasone and injections at L3 or below will contain 1,5 ml lidocaine 2% and 40mg methylprednisolone acetate in accordance with current Dutch anesthesiologic guidelines for usual care.
  Other Names: Transforaminal Epidural Steroid Injection

SUMMARY:
Rationale: Treatment with transforaminal epidural injections is part of usual care in patients suffering from lumbar radiculopathy. However, not all patients experience a satisfactory result from this treatment and it is unclear what percentage of patients responds well and if any clinical or radiological factors exist that predict a positive response.

Objectives:

Primary: to develop a model based on demographic, clinical and radiological parameters for prediction of treatment success after TEI

Secondary: to estimate the short-term efficacy of TEI in patients with LDH and spinal stenosis based on pain, functionality and perceived recovery scores, to determine the correlation between clinical and radiological baseline parameters and physical and psychological patient outcome measures, to determine the rate of additional injections and rate of surgery after treatment with TEI, to determine the short-term (cost)effectiveness of TEI on physical and psychological patient outcome measures, and to determine the rate of complications associated with TEI

Study design: Prospective cohort study

Study population: Patients that are scheduled for TEI as part of usual care suffering from a new episode of lumbar radiculopathy

Main study parameters/endpoints: leg and back pain scores at baseline, 30 minutes, 2 and 6 weeks after treatment. ODI, HADS, Quality of Life and PCI at baseline, 2 and 6 weeks after treatment. Perceived recovery at 2 and 6 weeks after treatment. Usage of healthcare at baseline, 2 and 6 weeks after treatment.

DETAILED DESCRIPTION:
Data collection schedule Baseline Weeks of follow-up 30 min. Day 4 Week 2 Week 6 Demographic data ✓ NRS leg pain ✓ ✓ ✓ ✓ NRS back pain ✓ ✓ ✓ ✓ ODI ✓ ✓ ✓ HADS ✓ ✓ ✓ QoL VAS ✓ ✓ ✓ PCI ✓ ✓ ✓ Likert score ✓ ✓ Adjuvant therapy ✓ ✓ ✓ TEI data ✓ ✓

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral lumbar radiculopathy secondary to LDH or one-level spinal stenosis
* Diagnosis supported by magnetic resonance imaging (MRI) findings
* Scheduled appointment for TEI
* Access to e-mail
* Signed informed consent

Exclusion Criteria:

* Diagnosis of unilateral lumbar radiculopathy secondary to LDH or one-level spinal stenosis
* Age under 18 years
* Severe multisegmental spinal disease
* Anatomical abnormalities that may complicate the procedure technically (e.g. severe scoliosis)
* Active malignancy or infectious disease
* Use of immunosuppressive drugs
* Use of systemic corticosteroids in preceding 3 months
* Previous treatment with TEI for current episode of lumbar radiculopathy
* History of lower back surgery at the same lumbar level
* Circumstances that prevent treatment with TEI (e.g. use of anticoagulants that cannot be temporarily discontinued, allergy against steroids or local anaesthetic)
* Pregnancy
* Major language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from lumbar radiculopathy due to lumbar disc herniation or spinal stenosis that have a scheduled appointment for treatment with TEI are screened to be candidates for this study. If the patient fulfills the inclusion and exclusion criteria the patient can participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale Leg Pain | 2 weeks
  The NRS score for leg pain

SECONDARY OUTCOMES:
Numerical Rating Scale Leg Pain | 30 minutes after treatment
  The NRS score for leg pain
Numerical Rating Scale Leg Pain | 6 weeks
  The NRS score for leg pain
Numerical Rating Scale Back Pain | 30 minutes after treatment
  The NRS score for back pain
Numerical Rating Scale Back Pain | 2 weeks
  The NRS score for back pain
Numerical Rating Scale Back Pain | 6 weeks
  The NRS score for back pain
Oswestry Disability Index | 2 weeks
  The ODI score for functionality
Oswestry Disability Index | 6 weeks
  The ODI score for functionality
Global Perceived Effect | 2 weeks
  The degree of patient satisfaction from experienced recovery on a Likert scale
Global Perceived Effect | 6 weeks
  The degree of patient satisfaction from experienced recovery on a Likert scale
Hospital Anxiety and Depression Scale | 2 weeks
  The HADS score for assessment of anxiety and depression
Hospital Anxiety and Depression Scale | 6 weeks
  The HADS score for assessment of anxiety and depression
Pain Coping Inventory | 2 weeks
  Assessment of the pain coping mechanisms of the patient
Pain Coping Inventory | 6 weeks
  Assessment of the pain coping mechanisms of the patient
Visual Analogue Scale Quality of Life | 2 weeks
  The VAS for assessment of Quality of Life
Visual Analogue Scale Quality of Life | 6 weeks
  The VAS for assessment of Quality of Life
Use of pain medication and physical therapy | 2 weeks
  Use of pain medication and physical therapy
Use of pain medication and physical therapy | 6 weeks
  Use of pain medication and physical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carmen LA Vleggeert-Lankamp, MD, PhD, Principal Investigator — Leiden University Medical Centre / Spaarne Gasthuis
Locations (1):
- Spaarne Gasthuis, Haarlem, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vroomen PC, de Krom MC, Knottnerus JA. Predicting the outcome of sciatica at short-term follow-up. Br J Gen Pract. 2002 Feb;52(475):119-23. PMID 11887877
- [Background] Sencan S, Celenlioglu AE, Asadov R, Gunduz OH. Predictive factors for treatment success of transforaminal epidural steroid injection in lumbar disc herniation-induced sciatica. Turk J Med Sci. 2020 Feb 13;50(1):126-131. doi: 10.3906/sag-1908-167. PMID 31742372
- [Background] Billy GG, Lin J, Gao M, Chow MX. Predictive Factors of the Effectiveness of Caudal Epidural Steroid Injections in Managing Patients With Chronic Low Back Pain and Radiculopathy. Clin Spine Surg. 2017 Jul;30(6):E833-E838. doi: 10.1097/BSD.0000000000000454. PMID 27764056
- [Background] Lee JW, Kim SH, Lee IS, Choi JA, Choi JY, Hong SH, Kang HS. Therapeutic effect and outcome predictors of sciatica treated using transforaminal epidural steroid injection. AJR Am J Roentgenol. 2006 Dec;187(6):1427-31. doi: 10.2214/AJR.05.1727. PMID 17114531
- [Background] McCormick Z, Cushman D, Casey E, Garvan C, Kennedy DJ, Plastaras C. Factors associated with pain reduction after transforaminal epidural steroid injection for lumbosacral radicular pain. Arch Phys Med Rehabil. 2014 Dec;95(12):2350-6. doi: 10.1016/j.apmr.2014.07.404. Epub 2014 Aug 7. PMID 25108099
- [Background] Cyteval C, Fescquet N, Thomas E, Decoux E, Blotman F, Taourel P. Predictive factors of efficacy of periradicular corticosteroid injections for lumbar radiculopathy. AJNR Am J Neuroradiol. 2006 May;27(5):978-82. PMID 16687527
- [Derived] Verheijen EJA, van Haagen OBHAM, Bartels EC, van der Sloot K, van den Akker-van Marle ME, Steyerberg EW, Vleggeert-Lankamp CLA. Prediction of transforaminal epidural injection success in sciatica (POTEISS): a protocol for the development of a multivariable prediction model for outcome after transforaminal epidural steroid injection in patients with lumbar radicular pain due to disc herniation or stenosis. BMC Neurol. 2024 Aug 20;24(1):290. doi: 10.1186/s12883-024-03801-1. PMID 39164613